CLINICAL TRIAL: NCT05691400
Title: Phase IV Multi-arm Study of CDK4/6 Pharmacokinetics in Healthy Volunteers With Known CYP3A4*22 Genotype
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding was not secured
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UMCC 2022.106; HUM00220623 (Other: University Of Michigan)
Record Dates: First submitted 2023-01-10; First posted 2023-01-20 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: CYP3A4*22
MeSH Terms: interventions — palbociclib; ribociclib; Tablets; abemaciclib

STUDY DESIGN:
Intervention Model Description: arms are designated based off of genotype; however, treatment is the same for each arm
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CYP3A4*1/*1 (Experimental): This arm will include subjects with CYP3A4*1/*1 genotype. They will receive a single oral dose of each CDK4/6 inhibitor on separate days, with at least 6 days and no more than 30 days between each medication. All participants will receive the medications in the same order: Palbociclib, Ribociclib, Abemaciclib
  Ribociclib- 200 mg tablet Abemaciclib- 150 mg tablet Palbociclib-125 mg tablet
  PK sampling will be done at the time of drug administration and at different time points until 48 hours post administration.
  Interventions: Drug: Palbociclib 125Mg Tab; Drug: Ribociclib 200Mg Oral Tablet; Drug: Abemaciclib 150 MG Oral Tablet
- CYP3A4*1/*22 (Experimental): This arm will include subjects with CYP3A4*1/*22 genotype. They will receive a single oral dose of each CDK4/6 inhibitor on separate days, with at least 6 days and no more than 30 days between each medication. All participants will receive the medications in the same order: Palbociclib, Ribociclib, Abemaciclib
  Ribociclib- 200 mg tablet Abemaciclib- 150 mg tablet Palbociclib-125 mg tablet
  PK sampling will be done at the time of drug administration and at different time points until 48 hours post administration.
  Interventions: Drug: Palbociclib 125Mg Tab; Drug: Ribociclib 200Mg Oral Tablet; Drug: Abemaciclib 150 MG Oral Tablet
- CYP3A4*22/*22 (Experimental): This arm will include subjects with CYP3A4*22/*22 genotype. They will receive a single oral dose of each CDK4/6 inhibitor on separate days, with at least 6 days and no more than 30 days between each medication. All participants will receive the medications in the same order: Palbociclib, Ribociclib, Abemaciclib
  Ribociclib- 200 mg tablet Abemaciclib- 150 mg tablet Palbociclib-125 mg tablet
  PK sampling will be done at the time of drug administration and at different time points until 48 hours post administration.
  Interventions: Drug: Palbociclib 125Mg Tab; Drug: Ribociclib 200Mg Oral Tablet; Drug: Abemaciclib 150 MG Oral Tablet

INTERVENTIONS:
Drug: Palbociclib 125Mg Tab — 125 mg single dose
  Other Names: ibrance
Drug: Ribociclib 200Mg Oral Tablet — 200 mg single dose
  Other Names: kisqali
Drug: Abemaciclib 150 MG Oral Tablet — 150 mg single dose
  Other Names: verzenio

SUMMARY:
The objective of this study is to estimate the effect of CYP3A4*22 on the clearance and area under the plasma concentration-time curve of Palbociclib, Ribociclib, and Abemaciclib

ELIGIBILITY:
Inclusion Criteria:

1. MGI participant with genotype of interest (e.g., CYP3A4*1/*1, CYP3A4*1/*22, or CYP3A4*22/*22) and consented to recontact for future research
2. Age≥18
3. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Concurrent use of a moderate or strong inhibitor or inducer of CYP3A4, based on the current version of the Drug Interactions Flockhart Table™, available at this link or by google search: https://drug-interactions.medicine.iu.edu/MainTable.aspx
2. Carriers another variant known to affect CYP3A4 activity, particularly CYP3A4*20.
3. Active malignancy or other disease state that would affect the pharmacokinetics of CDK4/6 inhibitors or place the participant at particular risk of toxicity from a single dose of a CDK4/6 inhibitor, in the opinion of the study team
4. History of allergic reaction to CDK4/6 inhibitor
5. Pregnancy or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Effect of CYP3A4*22 on the Clearance of Palbociclib | 2 days after initiation of Palbocicblib treatment
  To determine the effect of CYP3A4*22 on the Clearance of Palbociclib when administered as a single dose to healthy volunteers.
Effect of CYP3A4*22 on the Clearance of Ribociclib | up to 32 days after initiation of Study drug
  To determine the effect of CYP3A4*22 on the Clearance of Ribociclib when administered as a single dose to healthy volunteers.
Effect of CYP3A4*22 on the CL of Abemaciclib | up to 62 days after initiation of Study drug
  To determine the effect of CYP3A4*22 on the Clearance of Abemaciclib when administered as a single dose to healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Hertz, Principal Investigator — University of Michigan Rogel Cancer Center

IPD SHARING:
Plan to Share IPD: No
will be sharing individual participant data with collaborators at Rochester for analysis only